CLINICAL TRIAL: NCT05608967
Title: PREHapp Study Protocol: Effect of a Prehabilitation Mobile Application Versus Standard of Care Before Colon Cancer Surgery: a Randomized Pilot Study
Brief Title: Effect of a Prehabilitation Mobile Application Versus Standard of Care Before Colon Cancer Surgery.
Acronym: PREHAPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Luis Sánchez Guillen, MD, Staff Colorectal Surgeon, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: PREHAPP
Record Dates: First submitted 2022-10-10; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Prehabilitation; mHealth; Usability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- G_PREHapp: Experimental group will follow a prehabilitation programme through the PREHapp platform
  Interventions: Device: PREHapp
- G_Control: Control group will follow a prehabilitation programme according to usual practice

INTERVENTIONS:
Device: PREHapp — Prehabilitation programme through the PREHapp platform
  Groups: G_PREHapp

SUMMARY:
Pilot study to evaluate the effect of prehabilitation programme through a mobile application PREHapp in colon cancer surgery. The objectives of this pilot study were to evaluate the usability of the PREHapp for people undergoing colon cancer surgery, estimate the effect of the app on functional recovery after surgery and to evaluate complications during the postoperative period after 4 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Diagnosis of resectable colon cancer with elective surgery.
* Participants have at least 2 weeks to their operation date.
* Agree to collaborate in the study and sign the informed consent

Exclusion Criteria:

* Diagnosis of unresectable colon cancer.
* Inability to follow the prehabilitation programme.
* Participants be able to understand written and spoken Spanish.
* Subjects with previous nutritional supplements.
* Pre-anesthetic evaluation with results, according to the classification of the American Society of Anesthesiologists (ASA) IV or V.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is made up of patients scheduled for colon surgery due to malignant pathology at the General Hospital of Elche. Patients must be 18 years of age or older, have an Android smartphone, and accept the prehabilitation program.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Usability | 2 year
  Evaluate the usability of PREHapp with the System Usability Scale (SUS). The SUS is a reliable and valid 10-statement usability scale suitable to assess a wide range of eHealth technologies. The total SUS score ranges from 0 to 100, and higher scores reflect higher usability. An SUS score of at least 62.7 was considered acceptable, and 68 or above was regarded as above average in terms of usability quality

SECONDARY OUTCOMES:
Functional recovery | 2 year
  Estimate the effect of the prehabilitation with app on functional recovery measured with the 6-minute walk test.
Complications | 2 year
  Evaluate complications during the postoperative period after 4 weeks of follow-up: clavien-dindo classification

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No